CLINICAL TRIAL: NCT06515275
Title: Video-Supported Medication Education for Women Undergoing In Vitro Fertilization (IVF): Quality of Life and Psychosocial Effects
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Principal Investigator, Merve Coskun, Assistant Professor, Acibadem University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2024-8/313
Record Dates: First submitted 2024-07-17; First posted 2024-07-23 (Actual); Last update posted 2025-02-04 (Actual); Status verified 2025-01

CONDITIONS: Infertility; In Vitro Fertilization; Psychosocial Support Systems; Quality of Life; Health Education
MeSH Terms: conditions — Infertility; Health Education

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Randomized Controlled Experimental Design
Who Masked: Participant
Masking Description: In the single-blind method, subjects do not know which of the experimental or control groups they were selected and therefore which method was applied to them. The researcher knows the subjects selected for the experimental and control groups, and therefore which method was applied to which subjects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Participants will complete a demographic and treatment-related questionnaire. Prior to starting ovulation induction, they will complete the SCREENIVF, STAI, and FertiQol scales. On the first day of ovulation induction, participants will receive face-to-face and video-assisted education on prescribed medications, covering purpose, dose, administration, injection technique, timing, effects, and side effects. After follicle tracking confirms readiness for egg retrieval, participants will receive individual education on the ovulation-triggering medication, followed by QR code-linked educational videos specific to this medication. Post-oocyte aspiration, once sedation effects wear off, participants will complete the SCREENIVF, STAI, and FertiQol scales, along with an Education Satisfaction Evaluation Form.
  Interventions: Other: Education via video (QR code links)
- Control Group (No Intervention): Participants will complete a demographic and treatment-related questionnaire. Before starting ovulation induction, they will complete the SCREENIVF, STAI, and FertiQol scales. On the first day of ovulation induction, participants will receive face-to-face education on medication use, covering purpose, dose, administration, injection technique, timing, effects, and side effects. After ovulation induction, follicle tracking will occur. Upon readiness for egg retrieval, participants will receive individual education on the medication to trigger ovulation. After oocyte aspiration and recovery from sedation, participants will complete the SCREENIVF, STAI, and FertiQol scales, plus an Education Satisfaction Evaluation Form. Control group participants seeking continued treatment after a failed cycle will receive post-study access to video-assisted medication education via QR codes.

INTERVENTIONS:
Other: Education via video (QR code links) — Video education on self-administered medications for women undergoing IVF treatment
  Arms: Experimental Group

SUMMARY:
Reproductive health problems, particularly infertility, affect 48 million couples globally, ranking as the fifth most serious global obstacle for women. Infertility can lead to significant psychosocial effects, including stress, anxiety, and depression, with women experiencing these impacts more severely than men. In vitro fertilization (IVF) offers a solution but comes with emotional, physical, and psychosocial challenges, particularly for women, who often experience fatigue, headaches, weight gain, and stress. Effective support mechanisms, such as information and education, are crucial in improving the IVF experience. Video-assisted educational programs have shown promise in enhancing knowledge and reducing stress during IVF treatment. However, there is a lack of studies evaluating their impact on the quality of life and psychosocial status of women undergoing IVF. This study aims to examine the effect of video-supported training on drug use, quality of life, and psychosocial status of women during IVF treatment, hypothesizing that it will improve quality of life, increase emotional capacity, and reduce anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Being female
* Undergoing infertility treatment
* Aged 18-49 years
* Owning a tablet, smartphone, or similar device
* Having internet access
* Undergoing IVF treatment for the first time

Exclusion Criteria:

* Previously received controlled ovarian stimulation treatment
* Patients undergoing frozen embryo transfer
* No internet access
* Refusal to participate in the IVF medication teaching session

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2024-07-11 (Actual); Primary Completion 2025-02-11 (Estimated); Study Completion 2025-07-15 (Estimated)

PRIMARY OUTCOMES:
Introductory Information Form | to both groups before the intervention
  A 28-question form designed by researchers to gather sociodemographic, general health, obstetric, and gynecological history of the participants.
Screening Tool on Distress in Fertility Treatment's (SCREENIVF) | to both groups before the intervention and after oocyte aspiration (OPU)
  A tool recommended by ESHRE to assess psychosocial risk factors in individuals undergoing infertility treatment. The Turkish version consists of 28 items measuring anxiety, social support, helplessness, acceptance, and depression.
Fertility quality of life tool (FertiQoL) | to both groups before the intervention and after oocyte aspiration (OPU)
  A 36-item scale developed by Boivin et al. (2011) to assess the quality of life in individuals with fertility problems. The Turkish version was validated by Dural et al. (2016).
State-Trait Anxiety Inventory (STAI) | to both groups before the intervention and after oocyte aspiration (OPU)
  A 40-item inventory developed by Spielberger et al. (1970) and adapted to Turkish by Öner and Le Compte (1983). The inventory measures situational anxiety (20 items) and trait anxiety (20 items).
Education Satisfaction Evaluation Form | to both groups after oocyte aspiration (OPU)
  A form developed by researchers to assess satisfaction with medication education. It uses a 0-10 scale, with higher scores indicating greater satisfaction. The form for the experimental group will also record video viewing behavior.

CONTACTS AND LOCATIONS:
Locations (1):
- Merve Coşkun, Ataşehir, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] European Society of Human Reproduction and Embryology (ESHRE). (2021, August). Factsheet on infertility - prevalence, treatment and fertility decline in Europe.
- [Background] Gameiro S, Finnigan A. Long-term adjustment to unmet parenthood goals following ART: a systematic review and meta-analysis. Hum Reprod Update. 2017 May 1;23(3):322-337. doi: 10.1093/humupd/dmx001. PMID 28164236
- [Background] Ahmadi SM, Shahverdi J, Rezaei M, Bakhtiari M, Sadeghi K, Veisy F, Shahverdi M. The Effect of Behavioral Couple Therapy on the Improvement of Mental Health and Reduction of Marital Conflict in Infertile Couples in Kermanshah: A Randomized Controlled Trial (RCT). J Reprod Infertil. 2019 Jan-Mar;20(1):16-23. PMID 30859078
- [Background] Barnack-Tavlaris, J. L. (2019). Women's Experiences of Infertility. In J. C. C. Jane M. Ussher, Janette Perz (Ed.), Routledge International Handbook of Women's Sexual and Reproductive Health (pp. 205-220): Routledge.
- [Background] Bakhtiyar K, Beiranvand R, Ardalan A, Changaee F, Almasian M, Badrizadeh A, Bastami F, Ebrahimzadeh F. An investigation of the effects of infertility on Women's quality of life: a case-control study. BMC Womens Health. 2019 Sep 4;19(1):114. doi: 10.1186/s12905-019-0805-3. PMID 31484531
- [Background] Yassa, M., Arslan, E., & Gulbahar, D. S. (2019). Effects of infertility treatment on anxiety and depression levels. Cukurova Medical Journal, 44(2), 410-415.
- [Background] Gameiro S, Boivin J, Dancet E, de Klerk C, Emery M, Lewis-Jones C, Thorn P, Van den Broeck U, Venetis C, Verhaak CM, Wischmann T, Vermeulen N. ESHRE guideline: routine psychosocial care in infertility and medically assisted reproduction-a guide for fertility staff. Hum Reprod. 2015 Nov;30(11):2476-85. doi: 10.1093/humrep/dev177. Epub 2015 Sep 7. PMID 26345684
- [Background] LoGiudice JA, Massaro J. The impact of complementary therapies on psychosocial factors in women undergoing in vitro fertilization (IVF): A systematic literature review. Appl Nurs Res. 2018 Feb;39:220-228. doi: 10.1016/j.apnr.2017.11.025. Epub 2017 Nov 21. PMID 29422163
- [Background] Pasch LA, Holley SR, Bleil ME, Shehab D, Katz PP, Adler NE. Addressing the needs of fertility treatment patients and their partners: are they informed of and do they receive mental health services? Fertil Steril. 2016 Jul;106(1):209-215.e2. doi: 10.1016/j.fertnstert.2016.03.006. Epub 2016 Mar 24. PMID 27018159
- [Background] Vause TDR, Allison DJ, Vause T, Tekok-Kilic A, Ditor DS, Min JK. Comparison of a Web-Based Teaching Tool and Traditional Didactic Learning for In Vitro Fertilization Patients: A Preliminary Randomized Controlled Trial. J Obstet Gynaecol Can. 2018 May;40(5):588-594. doi: 10.1016/j.jogc.2017.08.029. Epub 2017 Oct 17. PMID 29054507
- [Background] Jones CA, Mehta C, Zwingerman R, Liu KE. Fertility patients' use and perceptions of online fertility educational material. Fertil Res Pract. 2020 Jul 18;6:11. doi: 10.1186/s40738-020-00083-2. eCollection 2020. PMID 32695432
- [Background] Mills R, Ensinger M, Callanan N, Haga SB. Development and Initial Assessment of a Patient Education Video about Pharmacogenetics. J Pers Med. 2017 May 25;7(2):4. doi: 10.3390/jpm7020004. PMID 28587070
- [Background] Park J, Son W, Park KS, Kang DH, Lee J, Oh CW, Kwon OK, Kim T, Kim CH. Educational and interactive informed consent process for treatment of unruptured intracranial aneurysms. J Neurosurg. 2017 Mar;126(3):825-830. doi: 10.3171/2016.2.JNS151830. Epub 2016 May 6. PMID 27153169
- [Background] Winter M, Kam J, Nalavenkata S, Hardy E, Handmer M, Ainsworth H, Lee WG, Louie-Johnsun M. The use of portable video media vs standard verbal communication in the urological consent process: a multicentre, randomised controlled, crossover trial. BJU Int. 2016 Nov;118(5):823-828. doi: 10.1111/bju.13595. Epub 2016 Aug 25. PMID 27440499
- [Background] Bernard AL, Barbour AK, Meernik C, Madeira JL, Lindheim SR, Goodman LR. The impact of an interactive multimedia educational platform on patient comprehension and anxiety during fertility treatment: a randomized controlled trial. F S Rep. 2022 May 22;3(3):214-222. doi: 10.1016/j.xfre.2022.05.006. eCollection 2022 Sep. PMID 36212557
- [Background] Boivin J, Takefman J, Braverman A. The fertility quality of life (FertiQoL) tool: development and general psychometric properties. Hum Reprod. 2011 Aug;26(8):2084-91. doi: 10.1093/humrep/der171. Epub 2011 Jun 10. PMID 21665875
- [Background] Verhaak CM, Lintsen AM, Evers AW, Braat DD. Who is at risk of emotional problems and how do you know? Screening of women going for IVF treatment. Hum Reprod. 2010 May;25(5):1234-40. doi: 10.1093/humrep/deq054. Epub 2010 Mar 13. PMID 20228392